CLINICAL TRIAL: NCT01044095
Title: Evaluation of In Vitro Cross-Reactivity With Avian Influenza H5N1 Virus in Healthy Volunteers Vaccinated With a Prime Boost Regimen of Seasonal Influenza Vaccine
Brief Title: Study of Seasonal Influenza Vaccine Against H5N1 Avian Influenza Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WRAIR1525; HSRRB No. A-15223 (Other: Human Subjects Research Review Board)
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Influenza
Keywords: seasonal influenza vaccine; avian influenza H5N1; cross reactivity; prime boost
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Autologous prime boost regimen 1 (Active Comparator): FluMist® live intranasal vaccine (LAIV) 0.2mL (0.1mL per nostril): 2 doses separated by 8 weeks (+/- 7 days)
  Interventions: Biological: FluMist® live, attenuated, intranasal seasonal influenza vaccine
- Autologous prime boost regimen 2 (Active Comparator): Fluzone® inactivated seasonal influenza virus vaccine intramuscularly: 2 doses separated by 8 weeks (+7 days)
  Interventions: Biological: Fluzone® inactivated influenza virus vaccine
- Heterologous prime boost regimen 1 (Experimental): FluMist® live, intranasal vaccine single dose, followed by Fluzone® inactivated influenza virus vaccine 8 weeks (+/-7 days) later
  Interventions: Biological: FluMist® live, attenuated, intranasal seasonal influenza vaccine; Biological: Fluzone® inactivated influenza virus vaccine
- Heterologous prime boost regimen 2 (Experimental): Fluzone® inactivated seasonal influenza virus vaccine single dose, followed by FluMist® live, intranasal seasonal influenza vaccine 0.2mL 8 weeks (+/- 7 days) later
  Interventions: Biological: FluMist® live, attenuated, intranasal seasonal influenza vaccine; Biological: Fluzone® inactivated influenza virus vaccine

INTERVENTIONS:
Biological: FluMist® live, attenuated, intranasal seasonal influenza vaccine — FluMist® live, attenuated, intranasal seasonal influenza vaccine 0.2mL (0.1mL per nostril)
  Arms: Autologous prime boost regimen 1; Heterologous prime boost regimen 1; Heterologous prime boost regimen 2
Biological: Fluzone® inactivated influenza virus vaccine — Fluzone® inactivated influenza virus vaccine 0.5mL intramuscularly
  Arms: Autologous prime boost regimen 2; Heterologous prime boost regimen 1; Heterologous prime boost regimen 2

SUMMARY:
This will be a randomized, open-label, pilot feasibility study of four 2-dose vaccine regimens in healthy volunteers using two commercially available seasonal influenza vaccines to compare immune responses and in vitro cross-reactivity against H5N1. Vaccine doses will be spaced by approximately 8 weeks to allow for optimal prime boost conditions. Humoral, cellular and secretory immune responses will be measured 2 and 4 weeks after each vaccine dose and compared with baseline values.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-49 years.
2. Healthy as determined by the PI or designate
3. Willing to give informed consent.
4. Willing to attend follow-up appointments and undergo study procedures.
5. US passport holder residing in Bangkok
6. If military, have a letter of approval for participation from the chain of command (Unit Commander).

Exclusion Criteria:

1. History of hypersensitivity to eggs, egg proteins, gentamicin, gelatin or arginine.
2. Severe or life-threatening reaction to any previous vaccine.
3. History of chronic respiratory illness, including asthma and sinusitis.
4. History of heart disease
5. History of kidney disease
6. Metabolic disease such as diabetes
7. Immunocompromised as determined by the PI, or a household contact of an immunocompromised individual.
8. History of Guillain-Barre syndrome.
9. Blood disease including sickle cell disease and/or bleeding tendency (by history or based on medical records).
10. Any influenza vaccination within the previous 6 months, or any other vaccine within 30 days of either dose of influenza vaccine.
11. Pregnant woman or nursing mother or unwilling to use reliable contraception during the study period until the final day of follow-up.
12. Blood donation within the preceding 3 months, or screening hemoglobin value of <12.5 g/dl.
13. Receipt of blood products including immunoglobulins within the preceding 3 months.
14. Receiving any of the following therapies: aspirin, warfarin, theophylline, phenytoin, aminopyrine, immunosuppressive drugs,
15. Receipt of any antiviral agents within 48 hours of vaccine administration.
16. HIV positive on screening blood tests.
17. Any other condition that in the opinion of the study investigator warrants exclusion from the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
antibody titers | 12 weeks

SECONDARY OUTCOMES:
safety of 2 doses of seasonal influenza vaccine in healthy adults | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Delia B Bethell, BM BCh, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand
Locations (1):
- United States Embassy Medical Unit, Bangkok, Thailand

REFERENCES:
- [Result] Bethell D, Saunders D, Jongkaewwattana A, Kramyu J, Thitithayanont A, Wiboon-ut S, Yongvanitchit K, Limsalakpetch A, Kum-Arb U, Uthaimongkol N, Garcia JM, Timmermans AE, Peiris M, Thomas S, Engering A, Jarman RG, Mongkolsirichaikul D, Mason C, Khemnu N, Tyner SD, Fukuda MM, Walsh DS, Pichyangkul S. Evaluation of in vitro cross-reactivity to avian H5N1 and pandemic H1N1 2009 influenza following prime boost regimens of seasonal influenza vaccination in healthy human subjects: a randomised trial. PLoS One. 2013;8(3):e59674. doi: 10.1371/journal.pone.0059674. Epub 2013 Mar 26. PMID 23555741
- See also: Related Info — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0059674